CLINICAL TRIAL: NCT00744263
Title: A Phase 4, Randomized, Placebo-Controlled Clinical Trial of 13-valent Pneumococcal Conjugate Vaccine Efficacy in Prevention of Vaccine-Serotype Pneumococcal Community-Acquired Pneumonia and Invasive Pneumococcal Disease
Brief Title: Study Evaluating the Effiacy of a 13-Valent Pneumococcal Conjugate Vaccine (13vPnC) in Adults
Acronym: CAPITA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 6115A1-3006; B1851025
Record Dates: First submitted 2008-08-27; First posted 2008-08-29 (Estimated); Results first posted 2014-10-06 (Estimated); Last update posted 2014-10-06 (Estimated); Status verified 2014-10

CONDITIONS: Pneumonia, Pneumococcal; Pneumococcal Infections; 13-valent Pneumococcal Vaccine
MeSH Terms: conditions — Pneumonia, Pneumococcal; Pneumococcal Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Biological: VACCINE: placebo
- 13-valent pneumococcal conjugate vaccine (Experimental)
  Interventions: Biological: VACCINE: 13-valent pneumococcal conjugate vaccine

INTERVENTIONS:
Biological: VACCINE: placebo — 0.5 mL, single intra-muscular injection
  Arms: Placebo
Biological: VACCINE: 13-valent pneumococcal conjugate vaccine — 0.5 mL, single intra-muscular injection
  Other Names: 13vPnC
  Arms: 13-valent pneumococcal conjugate vaccine

SUMMARY:
The purpose of this study is to assess the efficacy of 13-valent pneumococcal conjugate vaccine in the prevention of the first episode of vaccine-type pneumococcal community-acquired pneumonia in adults.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults aged 65 years or older on the day of vaccination and able to fulfill study requirements.

Exclusion Criteria:

* Previous vaccination with any licensed or experimental pneumococcal vaccine
* Residence in a nursing home, long-term care facility, or similar facility
* Known hypersensitivity to vaccination
* Immune deficiency or suppression

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 84496 (Actual)
Dates: Start 2008-09; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (98):
- Netherlands (98):
  - Pfizer Investigational Site, Tilburg, North Brabant
  - Pfizer Investigational Site, Abbekerk
  - Pfizer Investigational Site, Alkmaar
  - Pfizer Investigational Site, Almelo
  - Pfizer Investigational Site, Almere Stad
  - Pfizer Investigational Site, Alphen aan den Rijn
  - Pfizer Investigational Site, Amersfoort
  - Pfizer Investigational Site, Amstelveen
  - Pfizer Investigational Site, Amsterdam
  - Pfizer Investigational Site, Apeldoorn
  - Pfizer Investigational Site, Arnhem
  - Pfizer Investigational Site, Assen
  - Pfizer Investigational Site, Baarle-Nassau
  - Pfizer Investigational Site, Baarn
  - Pfizer Investigational Site, Bedum
  - Pfizer Investigational Site, Bennebroek
  - Pfizer Investigational Site, Bergen op Zoom
  - Pfizer Investigational Site, Berkel-Enschot
  - Pfizer Investigational Site, Berkhout
  - Pfizer Investigational Site, Bilthoven
  - Pfizer Investigational Site, Blaricum
  - Pfizer Investigational Site, Breda
  - Pfizer Investigational Site, Brunssum
  - Pfizer Investigational Site, Deventer
  - Pfizer Investigational Site, Dongen
  - Pfizer Investigational Site, Eelde
  - Pfizer Investigational Site, Eindhoven
  - Pfizer Investigational Site, Emmen
  - Pfizer Investigational Site, Enschede
  - Pfizer Investigational Site, Epe
  - Pfizer Investigational Site, Ettenleur
  - Pfizer Investigational Site, Fijnaart
  - Pfizer Investigational Site, Geldrop
  - Pfizer Investigational Site, Goirle
  - Pfizer Investigational Site, Gouda
  - Pfizer Investigational Site, Groningen
  - Pfizer Investigational Site, Grootebroek
  - Pfizer Investigational Site, Haarlem
  - Pfizer Investigational Site, Haren
  - Pfizer Investigational Site, Harmelen
  - Pfizer Investigational Site, Heerhugowaard
  - Pfizer Investigational Site, Heerlen
  - Pfizer Investigational Site, Heiloo
  - Pfizer Investigational Site, Helmond
  - Pfizer Investigational Site, Hengelo
  - Pfizer Investigational Site, Hilvarenbeek
  - Pfizer Investigational Site, Hilversum
  - Pfizer Investigational Site, Hoofddorp
  - Pfizer Investigational Site, Hoogezand
  - Pfizer Investigational Site, Hoorn
  - Pfizer Investigational Site, Houten
  - Pfizer Investigational Site, Kampen
  - Pfizer Investigational Site, Katwijk
  - Pfizer Investigational Site, Kerkrade
  - Pfizer Investigational Site, Leek
  - Pfizer Investigational Site, Leeuwarden
  - Pfizer Investigational Site, Leiden
  - Pfizer Investigational Site, Leiderdorp
  - Pfizer Investigational Site, Maarssen
  - Pfizer Investigational Site, Maastricht
  - Pfizer Investigational Site, Medemblik
  - Pfizer Investigational Site, Nieuwegein
  - Pfizer Investigational Site, Nijmegen
  - Pfizer Investigational Site, Noordwijk
  - Pfizer Investigational Site, Oldenzaal
  - Pfizer Investigational Site, Oosterhout
  - Pfizer Investigational Site, Peize
  - Pfizer Investigational Site, Rheden
  - Pfizer Investigational Site, Riel
  - Pfizer Investigational Site, Rijsbergen
  - Pfizer Investigational Site, Rijssen
  - Pfizer Investigational Site, Roden
  - Pfizer Investigational Site, Roermond
  - Pfizer Investigational Site, Roosendaal
  - Pfizer Investigational Site, Schoorl
  - Pfizer Investigational Site, Simpelveld
  - Pfizer Investigational Site, Sittard
  - Pfizer Investigational Site, Sleen
  - Pfizer Investigational Site, Soest
  - Pfizer Investigational Site, Son
  - Pfizer Investigational Site, Spaubeek
  - Pfizer Investigational Site, Steenbergen
  - Pfizer Investigational Site, Tiel
  - Pfizer Investigational Site, Tilburg
  - Pfizer Investigational Site, Uithoorn
  - Pfizer Investigational Site, Urmond
  - Pfizer Investigational Site, Utrecht
  - Pfizer Investigational Site, Veldhoven
  - Pfizer Investigational Site, Velp
  - Pfizer Investigational Site, Venlo
  - Pfizer Investigational Site, Waalwijk
  - Pfizer Investigational Site, Warmenhuizen
  - Pfizer Investigational Site, Weert
  - Pfizer Investigational Site, Woerden
  - Pfizer Investigational Site, Zeist
  - Pfizer Investigational Site, Zevenaar
  - Pfizer Investigational Site, Zutphen
  - Pfizer Investigational Site, Zwolle

REFERENCES:
- [Derived] Suaya JA, Jiang Q, Scott DA, Gruber WC, Webber C, Schmoele-Thoma B, Hall-Murray CK, Jodar L, Isturiz RE. Post hoc analysis of the efficacy of the 13-valent pneumococcal conjugate vaccine against vaccine-type community-acquired pneumonia in at-risk older adults. Vaccine. 2018 Mar 7;36(11):1477-1483. doi: 10.1016/j.vaccine.2018.01.049. Epub 2018 Feb 9. PMID 29429807
- [Derived] van Deursen AMM, van Houten MA, Webber C, Patton M, Scott DA, Patterson S, Sidhu M, Drews W, Gruber WC, Emini EA, Grobbee DE, Bonten MJM, Sanders EAM. Immunogenicity of the 13-Valent Pneumococcal Conjugate Vaccine in Older Adults With and Without Comorbidities in the Community-Acquired Pneumonia Immunization Trial in Adults (CAPiTA). Clin Infect Dis. 2017 Sep 1;65(5):787-795. doi: 10.1093/cid/cix419. PMID 29017280
- [Derived] Huijts SM, van Werkhoven CH, Bolkenbaas M, Grobbee DE, Bonten MJM. Post-hoc analysis of a randomized controlled trial: Diabetes mellitus modifies the efficacy of the 13-valent pneumococcal conjugate vaccine in elderly. Vaccine. 2017 Aug 3;35(34):4444-4449. doi: 10.1016/j.vaccine.2017.01.071. Epub 2017 Apr 12. PMID 28410813
- [Derived] Webber C, Patton M, Patterson S, Schmoele-Thoma B, Huijts SM, Bonten MJ; CAPiTA Study Group. Exploratory efficacy endpoints in the Community-Acquired Pneumonia Immunization Trial in Adults (CAPiTA). Vaccine. 2017 Mar 1;35(9):1266-1272. doi: 10.1016/j.vaccine.2017.01.032. Epub 2017 Feb 4. PMID 28173960
- [Derived] Bonten MJ, Huijts SM, Bolkenbaas M, Webber C, Patterson S, Gault S, van Werkhoven CH, van Deursen AM, Sanders EA, Verheij TJ, Patton M, McDonough A, Moradoghli-Haftvani A, Smith H, Mellelieu T, Pride MW, Crowther G, Schmoele-Thoma B, Scott DA, Jansen KU, Lobatto R, Oosterman B, Visser N, Caspers E, Smorenburg A, Emini EA, Gruber WC, Grobbee DE. Polysaccharide conjugate vaccine against pneumococcal pneumonia in adults. N Engl J Med. 2015 Mar 19;372(12):1114-25. doi: 10.1056/NEJMoa1408544. PMID 25785969
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=6115A1-3006&StudyName=Study%20Evaluating%20the%20effiacy%20of%20a%2013-Valent%20Pneumococcal%20Conjugate%20Vaccine%20%2813vPnC%29%20in%20Adults

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of 84496 participants who were randomized in this study, 2011 participants were included in the immunogenicity subset. Participants in the immunogenicity subset were analyzed for local reactions and systemic events as per planned analysis.
Groups:
- 13vPnC: Participants received a single 0.5 milliliter (mL) dose of 13-valent pneumococcal conjugate vaccine (13vPnC) intramuscular injection on Day 1.
- Placebo: Participants received placebo matched to a single dose of 13vPnC intramuscular injection on Day 1.
Period: Overall Study
Arm/Group | 13vPnC | Placebo
Started | 42240 | 42256
Completed | 37004 | 36936
Not Completed | 5236 | 5320
Not completed — Death | 3006 | 3005
Not completed — Lost to Follow-up | 2038 | 2135
Not completed — Withdrawal by Subject | 166 | 150
Not completed — Physician Decision | 20 | 23
Not completed — Protocol Violation | 3 | 5
Not completed — Adverse Event | 1 | 0
Not completed — Other | 2 | 2

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received study vaccine and who had any safety data.
Groups:
- Total: Total of all reporting groups
Arm/Group | 13vPnC | Placebo | Total
Number analyzed (Participants) | 42237 | 42255 | 84492
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.8 (5.7) | 72.8 (5.6) | 72.8 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18790 | 18454 | 37244
  Male | 23447 | 23801 | 47248

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With First Episode of Confirmed Vaccine-type Community-acquired Pneumonia (VT-CAP)
Description: CAP was defined based on clinical and radiological criteria. Microbiological criteria differentiate different categories of CAP. Clinical criteria: presence of 2 or more criteria from following: cough, production of purulent sputum/change in sputum character, temperature greater than (>) 38.0 degrees Celsius (C) or less than (<) 36.1 degrees C, auscultatory findings consistent with pneumonia including rales and/or evidence of pulmonary consolidation, leukocytosis (>10*10^9 white blood cells/liter or >15 percent (%) bands), C-reactive protein level >3 times upper limit of normal, hypoxemia with partial oxygen pressure <60 millimeter of mercury (mmHg). Radiological criteria: pneumonia confirmation by adjudication committee via lateral, posterior-anterior chest x-ray or anterior-posterior chest x-ray. Microbiological criteria: VT Streptococcus pneumonia culture from blood, pleural fluid or other sterile site and/or positive VT serotype-specific urinary antigen detection (SSUAD).
Time Frame: Baseline up to occurrence of first episode of VT-CAP, death, withdrawal of consent, loss to follow-up, participant request or end of case acquisition defined as accumulation of 130 VT cases (mean follow-up was 3.97 years)
Population: Per-protocol(PP) population: eligible participants who received study vaccine, 65 years or older, identified with CAP(pre-defined criteria) or had invasive pneumococcal disease(IPD); symptom onset at least 14 days after vaccination; immunocompetent at time of episode; no major protocol violations as determined by clinical scientist/medical monitor.
Measure: Number; unit: participants
Arm/Group | 13vPnC | Placebo
Number analyzed (Participants) | 42240 | 42256
participants | 49 | 90
Statistical Analysis 1: Comparison: 13vPnC vs Placebo; Vaccine efficacy against first event expressed as percentage. Vaccine efficacy = 1 - (proportion of participants who received 13vPnC with confirmed VT-CAP relative to those who received placebo). p-value and confidence intervals were derived using Clopper-Pearson method. The null hypothesis was vaccine efficacy = 0; Test type: Superiority or Other; p = 0.0006, Clopper-Pearson method; Vaccine Efficacy = 45.56, 95.2% CI 2-sided [21.82 to 62.49]

2. Secondary Outcome: Number of Participants With First Episode of Nonbacteremic/Noninvasive (NB/NI) Vaccine-type Community-acquired Pneumonia (VT-CAP)
Description: CAP was defined based on clinical and radiological criteria. Microbiological criteria differentiate different categories of CAP. Clinical criteria: presence of 2 or more criteria from following: cough, production of purulent sputum/change in sputum character, temperature >38.0 degrees C or <36.1 degrees C, auscultatory findings consistent with pneumonia including rales and/or evidence of pulmonary consolidation, leukocytosis (>10*10^9 white blood cells/liter or >15% bands), C-reactive protein level >3 times upper limit of normal, hypoxemia with partial oxygen pressure <60 mmHg. Radiological criteria: pneumonia confirmation by adjudication committee via lateral, posterior-anterior chest x-ray or anterior-posterior chest x-ray. Microbiological criteria: Confirmed VT pneumococcal CAP (by SSUAD) where a blood culture result was available and was negative and for which any other sterile culture results were negative for Streptococcus pneumoniae.
Time Frame: Baseline up to occurrence of first episode of NB/NI VT-CAP, death, withdrawal of consent, loss to follow-up, participant request or end of case acquisition defined as accumulation of 130 VT cases (mean follow-up was 3.97 years)
Population: PP population: eligible participants who received study vaccine, 65 years or older, identified with CAP (pre-defined criteria) or had IPD; symptom onset at least 14 days after vaccination; immunocompetent at time of episode; no major protocol violations as determined by clinical scientist/medical monitor.
Measure: Number; unit: participants
Arm/Group | 13vPnC | Placebo
Number analyzed (Participants) | 42240 | 42256
participants | 33 | 60
Statistical Analysis 1: Comparison: 13vPnC vs Placebo; Vaccine efficacy against first event expressed as percentage. Vaccine efficacy = 1-(proportion of participants who received 13vPnC with confirmed VT-CAP relative to those who received placebo). p-value and confidence intervals were derived using Clopper-Pearson method. The null hypothesis was vaccine efficacy = 0; Test type: Superiority or Other; p = 0.0067, Clopper-Pearson method; Vaccine Efficacy = 45.00, 95.2% CI 2-sided [14.21 to 65.31]

3. Secondary Outcome: Number of Participants With First Episodes of Vaccine-type Invasive Pneumococcal Disease (VT-IPD) Cases
Description: VT-IPD was defined as the presence of Streptococcus pneumoniae in a sterile site (blood, cerebrospinal fluid, pleural fluid, peritoneal fluid, pericardial fluid, surgical aspirate, bone, or joint fluid).
Time Frame: Baseline up to occurrence of first episode of VT-IPD, death, withdrawal of consent, loss to follow-up, participant request or end of case acquisition defined as accumulation of 130 VT cases (mean follow-up was 3.97 years)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | 13vPnC | Placebo
Number analyzed (Participants) | 42240 | 42256
participants | 7 | 28
Statistical Analysis 1: Comparison: 13vPnC vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0005, Clopper-Pearson method; Vaccine Efficacy = 75.00, 95% CI 2-sided [41.43 to 90.78]

4. Other Pre Specified Outcome: Percentage of Participants With Pre-specified Local Reactions Within 7 Days After Vaccination
Description: Local reactions were reported using electronic diary (e-diary). Redness and swelling scaled as Any (redness or swelling present); Absent (no or minimal); Mild (2.5 centimeter [cm] to 5.0 cm); Moderate (5.1 to 10.0 cm); Severe (>10.0 cm). Pain scaled as Any (pain present); Mild (did not interfere with activity); Moderate (interfered with activity); Severe (prevented daily activity). Limitation of arm movement scaled as Any (limitation present); Absent (no limitation of arm movement); Mild (some limitation of arm movement); Moderate (unable to move arm above head, but able to move arm above shoulder); Severe (unable to move arm above shoulder). Percentage of participants with local reactions were reported. Participants may be represented in more than 1 category.
Time Frame: Within 7 days after vaccination
Population: Immunogenicity subset included participants enrolled in the subset who received study vaccine, were able to complete e-diary and fulfilled other study procedures. Here 'N' (number of participants analyzed) signifies participants with known values for any local reaction and 'n' signifies participants with known values for specified local reaction.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC | Placebo
Number analyzed (Participants) | 917 | 867
percentage of participants
  Redness: Any (n = 886, 859) | 4.9 [3.5 to 6.5] | 1.2 [0.6 to 2.1]
  Redness: Mild (n = 886, 859) | 3.7 [2.6 to 5.2] | 0.8 [0.3 to 1.7]
  Redness: Moderate (n = 881, 859) | 1.7 [1.0 to 2.8] | 0.3 [0.1 to 1.0]
  Redness: Severe (n = 881, 859) | 0.5 [0.1 to 1.2] | 0.1 [0.0 to 0.6]
  Swelling: Any (n = 888, 859) | 6.8 [5.2 to 8.6] | 1.2 [0.6 to 2.1]
  Swelling: Mild (n = 888, 859) | 5.5 [4.1 to 7.2] | 0.7 [0.3 to 1.5]
  Swelling: Moderate (n = 884, 859) | 2.6 [1.7 to 3.9] | 0.6 [0.2 to 1.4]
  Swelling: Severe (n = 881, 859) | 0.1 [0.0 to 0.6] | 0.1 [0.0 to 0.6]
  Pain: Any (n = 914, 863) | 36.1 [33.0 to 39.3] | 6.1 [4.6 to 8.0]
  Pain: Mild (n = 913, 861) | 32.9 [29.8 to 36.0] | 5.6 [4.1 to 7.3]
  Pain: Moderate (n = 886, 860) | 7.7 [6.0 to 9.6] | 0.6 [0.2 to 1.4]
  Pain: Severe (n = 881, 860) | 0.3 [0.1 to 1.0] | 0.1 [0.0 to 0.6]
  Limitation of arm movement: Any (n = 891, 865) | 14.1 [11.9 to 16.6] | 3.2 [2.2 to 4.6]
  Limitation of arm movement: Mild (n = 888, 863) | 12.4 [10.3 to 14.7] | 2.5 [1.6 to 3.8]
  Limitation of arm movement: Moderate (n =883, 860) | 1.7 [1.0 to 2.8] | 0.5 [0.1 to 1.2]
  Limitation of arm movement: Severe (n = 882, 861) | 1.2 [0.6 to 2.2] | 0.7 [0.3 to 1.5]

5. Other Pre Specified Outcome: Percentage of Participants With Pre-specified Systemic Events Within 7 Days After Vaccination
Description: Systemic events (fever, fatigue, headache, chills, rash, vomiting, decreased appetite, diarrhea, new generalized muscle/joint pain [new muscle/joint pain], aggravated generalized muscle/joint pain [aggravated muscle/joint pain], use of medication to treat pain/fever) reported using an e-diary. Fever scaled as Absent(<38 degrees C); Mild(greater than or equal to [>=]38 to <38.5 degrees C); Moderate(>=38.5 to <39 degrees C); Severe(>=39 to less than or equal to [<=]40 degrees C); Potentially life threatening (>40 degrees C). Fatigue, headache, new/aggravated muscle/joint pain scaled as Mild(no interference); Moderate(some interference); Severe(prevented routine activity). Vomiting scaled as Mild(1-2 times in 24 hours [hrs]); Moderate(>2 times in 24 hrs); Severe(required intravenous hydration). Diarrhea scaled as Mild(2-3 loose stools in 24 hrs); Moderate(4-5 loose stools in 24 hrs); Severe(>=6 loose stools in 24 hrs). Percentage of participants with systemic events were reported.
Time Frame: Within 7 days after vaccination
Population: Immunogenicity subset. Participants may be represented in more than 1 category. Here 'N' (number of participants analyzed) signifies participants with known values for any systemic event and 'n' signifies participants with known values for specified systemic event.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC | Placebo
Number analyzed (Participants) | 918 | 907
percentage of participants
  Fever: >=38 to <38.5 degrees C (n = 883, 859) | 1.1 [0.5 to 2.1] | 0.6 [0.2 to 1.4]
  Fever: >=38.5 to <39 degrees C (n = 881, 859) | 0.6 [0.2 to 1.3] | 0.2 [0.0 to 0.8]
  Fever: >=39 to =<40 degrees C (n = 882, 859) | 0.7 [0.3 to 1.5] | 0.2 [0.0 to 0.8]
  Fever: >40 degrees C (n = 882, 860) | 0.8 [0.3 to 1.6] | 0.3 [0.1 to 1.0]
  Fatigue: Mild (n = 892, 871) | 13.8 [11.6 to 16.2] | 11.7 [9.7 to 14.0]
  Fatigue: Moderate (n = 886, 866) | 7.8 [6.1 to 9.8] | 6.2 [4.7 to 8.1]
  Fatigue: Severe (n = 883, 863) | 1.4 [0.7 to 2.4] | 0.9 [0.4 to 1.8]
  Headache: Mild (n = 891, 870) | 13.0 [10.9 to 15.4] | 13.1 [10.9 to 15.5]
  Headache: Moderate (n = 883, 868) | 5.2 [3.8 to 6.9] | 3.8 [2.6 to 5.3]
  Headache: Severe (n = 881, 861) | 0.6 [0.2 to 1.3] | 0.6 [0.2 to 1.3]
  Chills (n = 891, 866) | 9.4 [7.6 to 11.5] | 8.4 [6.7 to 10.5]
  Rash (n = 882, 860) | 3.3 [2.2 to 4.7] | 0.8 [0.3 to 1.7]
  Vomiting: Mild (n = 881, 860) | 0.0 [0.0 to 0.4] | 0.7 [0.3 to 1.5]
  Vomiting: Moderate (n =881, 860) | 0.1 [0.0 to 0.6] | 0.1 [0.0 to 0.6]
  Vomiting: Severe (n = 881, 860) | 0.2 [0.0 to 0.8] | 0.1 [0.0 to 0.6]
  Decreased appetite (n = 886, 865) | 5.3 [3.9 to 7.0] | 3.7 [2.5 to 5.2]
  Diarrhea: Mild (n = 887, 868) | 5.1 [3.7 to 6.7] | 7.7 [6.0 to 9.7]
  Diarrhea: Moderate (n = 882, 863) | 1.2 [0.6 to 2.2] | 1.0 [0.5 to 2.0]
  Diarrhea: Severe (n = 881, 862) | 0.7 [0.3 to 1.5] | 0.5 [0.1 to 1.2]
  New muscle pain: Mild (n = 894, 865) | 14.5 [12.3 to 17.0] | 6.7 [5.1 to 8.6]
  New muscle pain: Moderate (n = 886, 863) | 5.9 [4.4 to 7.6] | 2.8 [1.8 to 4.1]
  New muscle pain: Severe (n = 882, 860) | 0.7 [0.3 to 1.5] | 0.5 [0.1 to 1.2]
  Aggravated muscle pain: Mild (n = 886, 862) | 4.6 [3.3 to 6.2] | 1.9 [1.1 to 3.0]
  Aggravated muscle pain: Moderate (n = 885, 863) | 5.1 [3.7 to 6.7] | 2.8 [1.8 to 4.1]
  Aggravated muscle pain: Severe (n = 882, 860) | 0.7 [0.3 to 1.5] | 0.1 [0.0 to 0.6]
  New joint pain: Mild (n = 884, 862) | 5.0 [3.6 to 6.6] | 3.9 [2.7 to 5.5]
  New joint pain: Moderate (n = 883, 864) | 2.9 [1.9 to 4.3] | 2.2 [1.3 to 3.4]
  New joint pain: Severe (n = 882, 860) | 0.3 [0.1 to 1.0] | 0.3 [0.1 to 1.0]
  Aggravated joint pain: Mild (n = 883, 861) | 2.3 [1.4 to 3.5] | 1.7 [1.0 to 2.9]
  Aggravated joint pain: Moderate (n = 884, 862) | 3.2 [2.1 to 4.5] | 2.6 [1.6 to 3.8]
  Aggravated joint pain: Severe (n = 882, 860) | 0.3 [0.1 to 1.0] | 0.3 [0.1 to 1.0]
  Use of medication to treat pain (n = 887, 872) | 8.0 [6.3 to 10.0] | 6.2 [4.7 to 8.0]
  Use of medication to treat fever (n = 883, 863) | 3.2 [2.1 to 4.6] | 1.5 [0.8 to 2.6]

6. Other Pre Specified Outcome: Percentage of Participants Who Died
Description: Deaths collected throughout the case acquisition period were presented.
Time Frame: From signing of informed consent form up to case acquisition period defined as accumulation of 130 VT cases (mean follow-up was 3.97 years)
Population: Safety population included all participants who received study vaccine and who had any safety data.
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC | Placebo
Number analyzed (Participants) | 42237 | 42255
percentage of participants | 7.1 | 7.1
Statistical Analysis 1: Comparison: 13vPnC vs Placebo; Fisher exact test, 2-sided, was used to calculate the p-value for the difference between vaccine groups in percentages of participants; Test type: Superiority or Other; p = 0.979, Fisher Exact

7. Other Pre Specified Outcome: Percentage of Participants With Newly Diagnosed Chronic Medical Condition
Description: Percentage of participants with newly diagnosed chronic medical conditions (including autoimmune or neuroinflammatory disease) in the immunogenicity subset were reported as per planned analysis.
Time Frame: From 1 month after vaccination up to 6 months after vaccination
Population: Immunogenicity subset included participants enrolled in the subset who received study vaccine, were able to complete e-diary and fulfilled other study procedures.
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC | Placebo
Number analyzed (Participants) | 1006 | 1005
percentage of participants | 1.7 | 1.2
Statistical Analysis 1: Comparison: 13vPnC vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.455, Fisher Exact

ADVERSE EVENTS:
Time Frame: Safety set (SAEs: Day 1 up to 1 month after vaccination); Immunogenicity subset (SAEs:1 month up to 6 month after vaccination; Other AEs: Day 1 up to 1 month after vaccination; pre-specified local reactions, systemic events:up to 7 days after vaccination)
Description: SAEs were collected up to 1 month after vaccination for safety set. For immunogenicity subset, other AEs were collected up to 1 month after vaccination and SAEs collected from 1 month up to 6 months after vaccination. Deaths collected throughout case acquisition period but reported as SAE only during SAE collection periods as per planned analysis.
Groups:
- 13vPnC Safety Set: All Participants who received a single 0.5 milliliter (mL) dose of 13-valent pneumococcal conjugate vaccine (13vPnC) intramuscular injection on Day 1, were assessed for serious adverse events (SAEs) from vaccination up to 1 month after vaccination. Safety set included all participants who received study vaccine and who had any safety data.
- Placebo Safety Set: All participants who received placebo matched to a single dose of 13vPnC intramuscular injection on Day 1, were assessed for SAEs from vaccination up to 1 month after vaccination. Safety set included all participants who received study vaccine and who had any safety data.
- 13vPnC Immunogenicity Subset: Participants included in immunogenicity subset who received a single 0.5 mL dose of 13vPnC intramuscular injection on Day 1, were assessed for SAEs from 1 month after vaccination up to 6 months after vaccination and for Other adverse events (AEs) from vaccination up to 1 month after vaccination. Immunogenicity subset included participants enrolled in the subset who received study vaccine, were able to complete e-diary and fulfilled other study procedures.
- Placebo Immunogenicity Subset: Participants included in immunogenicity subset who received placebo matched to a single dose of 13vPnC intramuscular injection on Day 1, were assessed for SAEs from 1 month after vaccination up to 6 months after vaccination and for Other AEs from vaccination up to 1 month after vaccination. Immunogenicity subset included participants enrolled in the subset who received study vaccine, were able to complete e-diary and fulfilled other study procedures.
Arm/Group | 13vPnC Safety Set | Placebo Safety Set | 13vPnC Immunogenicity Subset | Placebo Immunogenicity Subset
Serious Adverse Events (participants affected / at risk) | 327/42237 | 314/42255 | 55/1006 | 48/1005
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 363/1006 | 315/1005
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 13vPnC Safety Set (N=42237) | Placebo Safety Set (N=42255) | 13vPnC Immunogenicity Subset (N=1006) | Placebo Immunogenicity Subset (N=1005)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 1 | 0
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 19 | 19 | 3 | 1
Atrial fibrillation (Cardiac disorders) | 13 | 9 | 3 | 1
Myocardial infarction (Cardiac disorders) | 12 | 6 | 0 | 1
Cardiac failure (Cardiac disorders) | 7 | 10 | 4 | 0
Atrial flutter (Cardiac disorders) | 5 | 2 | 0 | 0
Coronary artery disease (Cardiac disorders) | 3 | 4 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 2 | 3 | 1 | 0
Cardiac asthma (Cardiac disorders) | 2 | 3 | 0 | 0
Angina unstable (Cardiac disorders) | 2 | 2 | 0 | 0
Cardiac arrest (Cardiac disorders) | 2 | 1 | 0 | 1
Sick sinus syndrome (Cardiac disorders) | 1 | 2 | 0 | 0
Aortic valve stenosis (Cardiac disorders) | 1 | 1 | 1 | 0
Atrioventricular block (Cardiac disorders) | 1 | 1 | 0 | 0
Atrioventricular block complete (Cardiac disorders) | 1 | 1 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 1 | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 2 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0
Atrial tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1 | 0 | 0
Coronary artery dissection (Cardiac disorders) | 1 | 0 | 0 | 0
Left ventricular failure (Cardiac disorders) | 0 | 1 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0
Silent myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 1 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Retinal detachment (Eye disorders) | 1 | 1 | 0 | 0
Retinal artery occlusion (Eye disorders) | 1 | 0 | 0 | 0
Macular fibrosis (Eye disorders) | 0 | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 2 | 4 | 0 | 0
Constipation (Gastrointestinal disorders) | 4 | 1 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Duodenal perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastric perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Inguinal hernia, obstructive (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Subileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Varices oesophageal (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Large intestinal stenosis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 12 | 2 | 0 | 0
Chest pain (General disorders) | 5 | 1 | 0 | 0
Device dislocation (General disorders) | 2 | 0 | 1 | 0
Accidental death (General disorders) | 0 | 1 | 0 | 0
Death (General disorders) | 0 | 1 | 0 | 0
Device occlusion (General disorders) | 0 | 1 | 0 | 0
Hernia obstructive (General disorders) | 0 | 1 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0 | 0
Medical device complication (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 1 | 0
Sudden cardiac death (General disorders) | 1 | 0 | 0 | 0
Implant site fibrosis (General disorders) | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 2 | 2 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 2 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 2 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 2 | 0 | 0
Anaphylactic shock (Immune system disorders) | 0 | 1 | 0 | 1
Corneal graft rejection (Immune system disorders) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 14 | 6 | 4 | 1
Appendicitis (Infections and infestations) | 2 | 4 | 0 | 0
Device related infection (Infections and infestations) | 3 | 2 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 3 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 3 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 3 | 1 | 0
Pneumonia pneumococcal (Infections and infestations) | 1 | 2 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 1 | 0 | 0
Pneumonia legionella (Infections and infestations) | 1 | 1 | 0 | 0
Wound infection (Infections and infestations) | 0 | 2 | 2 | 1
Bronchiolitis (Infections and infestations) | 0 | 1 | 0 | 0
Cholangitis suppurative (Infections and infestations) | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0 | 0
Erysipelas (Infections and infestations) | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 0 | 0 | 0
Meningitis (Infections and infestations) | 1 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 1 | 0 | 0 | 0
Peritonsillar abscess (Infections and infestations) | 0 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0 | 0
Tuberculosis (Infections and infestations) | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Vestibular neuronitis (Infections and infestations) | 0 | 1 | 0 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Abdominal abscess (Infections and infestations) | 0 | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 5 | 4 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 3 | 3 | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 3 | 2 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 4 | 0 | 0
Brain contusion (Injury, poisoning and procedural complications) | 2 | 2 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 3 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 3 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 3 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 3 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Cardiac valve replacement complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Foreign body aspiration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Kidney contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Ligament injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Mental status changes postoperative (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Post laminectomy syndrome (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Procedural intestinal perforation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Tendon injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Urinary retention postoperative (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 1 | 0 | 0 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Finger deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Bone cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 22 | 16 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 | 7 | 0 | 2
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 6 | 2 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3 | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0
Bladder adenocarcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Hepatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Hypopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Malignant neoplasm of renal pelvis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Melanoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Oesophageal carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Bile duct adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Renal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 9 | 8 | 3 | 1
Cerebral infarction (Nervous system disorders) | 4 | 9 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 8 | 5 | 0 | 0
Syncope (Nervous system disorders) | 3 | 3 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 3 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 2 | 1 | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 2 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 2 | 0 | 0
Loss of consciousness (Nervous system disorders) | 1 | 1 | 0 | 0
Transient global amnesia (Nervous system disorders) | 0 | 2 | 0 | 0
Acute disseminated encephalomyelitis (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 1 | 0 | 0 | 0
Peroneal nerve palsy (Nervous system disorders) | 0 | 1 | 0 | 0
Radicular pain (Nervous system disorders) | 0 | 1 | 0 | 0
Radiculitis lumbosacral (Nervous system disorders) | 0 | 1 | 0 | 0
Trigeminal neuralgia (Nervous system disorders) | 1 | 0 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1 | 0
Peripheral nerve lesion (Nervous system disorders) | 0 | 0 | 0 | 1
Bipolar disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0 | 0
Calculus bladder (Renal and urinary disorders) | 2 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 2 | 0 | 1 | 0
Cystitis noninfective (Renal and urinary disorders) | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0 | 0
Ureteric stenosis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urethral stenosis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 2 | 1 | 1
Acquired phimosis (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Female genital tract fistula (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 13 | 8 | 2 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Alveolitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Circulatory collapse (Vascular disorders) | 3 | 2 | 1 | 0
Aortic aneurysm (Vascular disorders) | 2 | 1 | 2 | 0
Aortic aneurysm rupture (Vascular disorders) | 3 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0 | 1
Hypotension (Vascular disorders) | 2 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0 | 0
Intermittent claudication (Vascular disorders) | 0 | 1 | 2 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1 | 0 | 0
Temporal arteritis (Vascular disorders) | 1 | 0 | 0 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0 | 0 | 0
Malignant hypertension (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | 13vPnC Safety Set (N=0) | Placebo Safety Set (N=0) | 13vPnC Immunogenicity Subset (N=1006) | Placebo Immunogenicity Subset (N=1005)
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 0 | 5 | 0
Cataract (Eye disorders) | 0 | 0 | 1 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 0 | 1
Ocular hyperaemia (Eye disorders) | 0 | 0 | 1 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 3 | 5
Nausea (Gastrointestinal disorders) | 0 | 0 | 2 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Change of bowel habit (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Eructation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Injection site erythema (General disorders) | 0 | 0 | 30 | 0
Injection site pain (General disorders) | 0 | 0 | 18 | 2
Injection site pruritus (General disorders) | 0 | 0 | 10 | 0
Injection site swelling (General disorders) | 0 | 0 | 10 | 0
Malaise (General disorders) | 0 | 0 | 4 | 3
Fatigue (General disorders) | 0 | 0 | 2 | 4
Injection site haematoma (General disorders) | 0 | 0 | 1 | 2
Injection site exfoliation (General disorders) | 0 | 0 | 2 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 1
Chills (General disorders) | 0 | 0 | 1 | 0
Cyst (General disorders) | 0 | 0 | 1 | 0
Device breakage (General disorders) | 0 | 0 | 0 | 1
Ill-defined disorder (General disorders) | 0 | 0 | 1 | 0
Injection site rash (General disorders) | 0 | 0 | 1 | 0
Injection site reaction (General disorders) | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0
Vaccination site erythema (General disorders) | 0 | 0 | 1 | 0
Vessel puncture site haematoma (General disorders) | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 12 | 20
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 8 | 17
Cystitis (Infections and infestations) | 0 | 0 | 5 | 8
Gastroenteritis (Infections and infestations) | 0 | 0 | 4 | 9
Bronchitis (Infections and infestations) | 0 | 0 | 5 | 4
Influenza (Infections and infestations) | 0 | 0 | 4 | 5
Herpes zoster (Infections and infestations) | 0 | 0 | 2 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 3
Sinusitis (Infections and infestations) | 0 | 0 | 2 | 1
Fungal infection (Infections and infestations) | 0 | 0 | 2 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 1
Wound infection (Infections and infestations) | 0 | 0 | 0 | 2
Abscess oral (Infections and infestations) | 0 | 0 | 0 | 1
Enteritis infectious (Infections and infestations) | 0 | 0 | 1 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 1
Fungal skin infection (Infections and infestations) | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 1 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 1
Otitis media (Infections and infestations) | 0 | 0 | 1 | 0
Tinea barbae (Infections and infestations) | 0 | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Bone contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Face injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Periorbital contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
International normalised ratio decreased (Investigations) | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 3
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 5 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 3
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Inclusion body myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 7 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 3 | 3
Ageusia (Nervous system disorders) | 0 | 0 | 0 | 1
Aphonia (Nervous system disorders) | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 5 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Blood blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0
Peripheral coldness (Vascular disorders) | 0 | 0 | 0 | 1
Redness: Any (Skin and subcutaneous tissue disorders) | 0 | 0 | 43/886 | 10/859
Redness: Mild (Skin and subcutaneous tissue disorders) | 0 | 0 | 33/886 | 7/859
Redness: Moderate (Skin and subcutaneous tissue disorders) | 0 | 0 | 15/881 | 3/859
Redness: Severe (Skin and subcutaneous tissue disorders) | 0 | 0 | 4/881 | 1/859
Swelling: Any (Skin and subcutaneous tissue disorders) | 0 | 0 | 60/888 | 10/859
Swelling: Mild (Skin and subcutaneous tissue disorders) | 0 | 0 | 49/888 | 6/859
Swelling: Moderate (Skin and subcutaneous tissue disorders) | 0 | 0 | 23/884 | 5/859
Swelling: Severe (Skin and subcutaneous tissue disorders) | 0 | 0 | 1/881 | 1/859
Pain: Any (Skin and subcutaneous tissue disorders) | 0 | 0 | 330/914 | 53/863
Pain: Mild (Skin and subcutaneous tissue disorders) | 0 | 0 | 300/913 | 48/861
Pain: Moderate (Skin and subcutaneous tissue disorders) | 0 | 0 | 68/886 | 5/860
Pain: Severe (Skin and subcutaneous tissue disorders) | 0 | 0 | 3/881 | 1/860
Limitation of arm movement: Any (Skin and subcutaneous tissue disorders) | 0 | 0 | 126/891 | 28/865
Limitation of arm movement: Mild (Skin and subcutaneous tissue disorders) | 0 | 0 | 110/888 | 22/863
Limitation of arm movement: Moderate (Skin and subcutaneous tissue disorders) | 0 | 0 | 15/883 | 4/860
Limitation of arm movement: Severe (Skin and subcutaneous tissue disorders) | 0 | 0 | 11/882 | 6/861
Fever: >=38 to <38.5 degrees C (General disorders) | 0 | 0 | 10/883 | 5/859
Fever: >=38.5 to <39 degrees C (General disorders) | 0 | 0 | 5/881 | 2/859
Fever: >=39 to =<40 degrees C (General disorders) | 0 | 0 | 6/882 | 2/859
Fever: >40 degrees C (General disorders) | 0 | 0 | 7/882 | 3/860
Fatigue: Mild (General disorders) | 0 | 0 | 123/892 | 102/871
Fatigue: Moderate (General disorders) | 0 | 0 | 69/886 | 54/866
Fatigue: Severe (General disorders) | 0 | 0 | 12/883 | 8/863
Headache: Mild (General disorders) | 0 | 0 | 116/891 | 114/870
Headache: Moderate (General disorders) | 0 | 0 | 46/883 | 33/868
Headache: Severe (General disorders) | 0 | 0 | 5/881 | 5/861
Chills (General disorders) | 0 | 0 | 84/891 | 73/866
Rash (General disorders) | 0 | 0 | 29/882 | 7/860
Vomiting: Mild (General disorders) | 0 | 0 | 0/881 | 6/860
Vomiting: Moderate (General disorders) | 0 | 0 | 1/881 | 1/860
Vomiting: Severe (General disorders) | 0 | 0 | 2/881 | 1/860
Decreased appetite (General disorders) | 0 | 0 | 47/886 | 32/865
Diarrhea: Mild (General disorders) | 0 | 0 | 45/887 | 67/868
Diarrhea: Moderate (General disorders) | 0 | 0 | 11/882 | 9/863
Diarrhea: Severe (General disorders) | 0 | 0 | 6/881 | 4/862
New generalized muscle pain: Mild (General disorders) | 0 | 0 | 130/894 | 58/865
New generalized muscle pain: Moderate (General disorders) | 0 | 0 | 52/886 | 24/863
New generalized muscle pain: Severe (General disorders) | 0 | 0 | 6/882 | 4/860
Aggravated generalized muscle pain: Mild (General disorders) | 0 | 0 | 41/886 | 16/862
Aggravated generalized muscle pain: Moderate (General disorders) | 0 | 0 | 45/885 | 24/863
Aggravated generalized muscle pain: Severe (General disorders) | 0 | 0 | 6/882 | 1/860
New generalized joint pain: Mild (General disorders) | 0 | 0 | 44/884 | 34/862
New generalized joint pain: Moderate (General disorders) | 0 | 0 | 26/883 | 19/864
New generalized joint pain: Severe (General disorders) | 0 | 0 | 3/882 | 3/860
Aggravated generalized joint pain: Mild (General disorders) | 0 | 0 | 20/883 | 15/861
Aggravated generalized joint pain: Moderate (General disorders) | 0 | 0 | 28/884 | 22/862
Aggravated generalized joint pain: Severe (General disorders) | 0 | 0 | 3/882 | 3/860

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.